CLINICAL TRIAL: NCT01940770
Title: Specific Clinical Experience Investigation for Long-term Use of Bydureon Subcutaneous Injection 2 mg and Bydureon Subcutaneous Injection 2 mg PEN
Brief Title: Specific Clinical Experience Investigation for Long-term Use of Bydureon.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5551C00001; EUPAS18608 (Registry Identifier: ENCePP)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus(DM); Bydureon; Exenatide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To confirm the safety and efficacy of Bydureon in long-term use in Japanese patients with type 2 diabetes mellitus under actual drug use.

DETAILED DESCRIPTION:
To confirm the safety and efficacy of Bydureon (hereinafter referred to as Bydureon) in long-term use in Japanese patients with type 2 diabetes mellitus under actual drug use.

1. Primary Objective To confirm the safety profile in Japanese patients with type 2 diabetes mellitus receiving Bydureon under daily practices.
2. Secondary objective As the secondary objective of this S-CEI, the following items are to be investigated.

   * Frequencies of AEs related to cardiovascular events, hypoglycaemia, digestive symptoms, and injection site reaction.
   * Development of pancreatitis, renal impairment (especially acute renal failure), hypersensitivity reaction, and malignant tumour (especially thyroid tumour and pancreatic malignancy)
   * Safety in patients with mild or moderate renal impairment
   * Changes of weight, blood pressure, pulse rate, fasting blood sugar, fasting insulin, HbA1c, and blood lipids
   * Bydureon administration under daily practices focusing on the patient's demographics and clinical characteristics of diabetes mellitus (duration of diabetes mellitus, treatment duration, complications, Bydureon administration, etc)
   * Anti-exenatide antibody titer in AE cases (hypersensitivity, loss of control of blood sugar)

ELIGIBILITY:
Inclusion Criteria:

- The patients with type 2 diabetes mellitus who inadequately respond to sulfonylurea, biuguanides, and/or thiazolidines (monotherapy or combination use) in addition to diet and exercise.

Exclusion Criteria:

* No past history of hypersensitivity to the components of Bydureon.
* Not the patient with diabetic ketoacidosis, diabetic coma/ precoma, and/ or type 1 diabetes mellitus.
* Bydureon will not be administered to the patient in an emergency situation such as severe infection and operation.
* Not the patient with severe renal impairment, including those receiving dialysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with type 2 diabetes mellitus who will be given Bydureon for the first time and who inadequately respond to sulfonylurea, biuguanides, and/or thiazolidines (monotherapy or combination use) in addition to diet and exercise.
Sampling Method: Non-Probability Sample
Enrollment: 1137 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | 3 years
  Number of Adverse Drug Reactions

SECONDARY OUTCOMES:
Mean change of HbA1c | from baseline up to 3 years
  Change value of HbA1c from baseline as mean.
Mean change of weight | from baseline up to 3 years
  Change value of weight from baseline as mean.
Mean change of blood pressure | from baseline up to 3 years
  Change value of blood pressure from baseline as mean.
Mean change of lipid metabolism | from baseline up to 3 years
  Change value of lipid metabolism from baseline as mean.
Mean change of HbA1c | from baseline up to 3 years
  Change value of HbA1c from baseline as median.
Mean change of HbA1c | from baseline up to 3 years
  Change value of HbA1c from baseline as minimum.
Mean change of HbA1c | from baseline up to 3 years
  Change value of HbA1c from baseline as max.
Mean change of weight | from baseline up to 3 years
  Change value of weight from baseline as median.
Mean change of weight | from baseline up to 3 years
  Change value of weight from baseline as minimum.
Mean change of weight | from baseline up to 3 years
  Change value of weight from baseline as max.
Mean change of blood pressure | from baseline up to 3 years
  Change value of blood pressure from baseline as median.
Mean change of blood pressure | from baseline up to 3 years
  Change value of blood pressure from baseline as minimum.
Mean change of blood pressure | from baseline up to 3 years
  Change value of blood pressure from baseline as max.
Mean change of lipid metabolism | from baseline up to 3 years
  Change value of lipid metabolism from baseline as median.
Mean change of lipid metabolism | from baseline up to 3 years
  Change value of lipid metabolism from baseline as minimum.
Mean change of lipid metabolism | from baseline up to 3 years
  Change value of lipid metabolism from baseline as max.

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — Quality & Safety Compliance Office
Locations (47):
- Japan (47):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5551C00001&attachmentIdentifier=e0b68d9f-b1cc-4a28-ab50-d0860e405417&fileName=D5551C00001_redacted_CSR_Synopsis.PDF&versionIdentifier=